CLINICAL TRIAL: NCT00600808
Title: A Phase II/IIIa, Assessor Blinded (Partially Blinded), Randomised, Active-Controlled, Multicentre, Parallel-Group Study of the Safety, Efficacy and pk/pd of LB03002 Administered Weekly in Children With Growth Failure Due to GH Deficiency.
Brief Title: Sustained Release Formulation of Somatropin (rDNA Origin)for Injection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioPartners GmbH (Industry)
Collaborators: LG Life Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPLG-003
Record Dates: First submitted 2007-07-23; First posted 2008-01-25 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2007-07

CONDITIONS: Growth Hormone Deficiency
Keywords: SR-hGH, Pharmacokinetics, Pharmacodynamics
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: BPLG-003

SUMMARY:
Annualised height velocity after 12/24 months treatment and HV SDS height velocity after 12/24 months treatment expressed as number of standard deviations difference from the mean population height velocity for the appropriate gender and chronological age.

DETAILED DESCRIPTION:
To evaluate the safety, efficacy and pharmacokinetics/ pharmacodynamics of LB03002 in the treatment of growth failure in children with growth hormone deficiency (GHD) and to determine the dose for a subsequent phase IIIb BPLG-004 study

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of GHD as determined by two different GH provocation tests documenting deficient GH secretion, defined as a peak plasma GH level of less than 7 ng/mL and absence of any peak plasma GH level in the spontaneous growth hormone secretion above 7 ng/mL monitored 3 hours before the application of the pharmacological stimuli at least before one stimulation test.
* Pre-pubertal children (boys age: 4-10 years or girls: age 4-9 years) with primary (idiopathic) and secondary (organic) insufficiency of growth hormone secretion.
* Children with negative signs for intracranial tumour or tumour growth as confirmed with Computer tomography (CT) or magnetic resonance imaging (MRI) scan within 12 months prior to inclusion or within 6 months prior to inclusion of children with GH insufficiency occurred after treatment for any brain tumour. Such patients have to be at least 24 months into full clinical remission.
* No prior exposure to rhGH (GH-naïve)
* Height (HT) of at least 2.0 standard deviation (SD) (HT SDS ≤2.0) below the mean height for chronological age (CA) and sex according to the Standards of Prader et al15.
* Height Velocity (HV) of at least -1 SD (HV SDS ≤1) below the mean HV for CA and sex according to the Standards of Prader et al15.
* Baseline IGF-I level standardized for age and sex less than -1.0 SDS
* Bone age (BA) ≤9 years for boys and ≤ 8 years for girls,
* For children with multiple hormonal deficiencies, stabilized on replacement therapies for other pituitary axes (e.g. thyroid-stimulating hormone, adrenocorticotropic hormone/cortisol and vasopressin) for at least 3 months and 6 months for thyroid replacement therapy prior to enrolment for children with multiple hormonal deficiencies.
* Written informed consent of parent or legal guardian of subject.

Exclusion Criteria:

* The result of the 3 hours spontaneous GH peak is equal to, or above 7 ng/ml. The value of the peak GH level in case of repeated pharmacology test is below 7 ng/ml, whilst the 6 hours spontaneous peak GH is above this value,
* Any clinically significant abnormality likely to affect growth or the ability to evaluate growth, such as, but not limited to chronic diseases like renal insufficiency, diabetes mellitus and malnutrition (BMI must be above -2SD and below +2SD of mean BMI for the chronological age and sex, and albumin must be above lower limit of normal (LLN) of the central laboratory for a patient to be included), Chromosomal abnormalities and medical "syndromes", with the exception of holoprosencephaly/septo-optic dysplasia (Turner's syndrome, Laron syndrome, Noonan syndrome or absence of growth hormone receptors).
* Congenital abnormalities (causing skeletal abnormalities), Russell-Silver Syndrome, Skeletal dysplasias, Closed epiphyses,
* Other growth promoting medication such as anabolic steroids, with the exception of pituitary hormone replacement therapy, thyroxine, hydrocortisone and desmopressin (DDAVP) replacement therapies,
* Children requiring glucocorticoid therapy (e.g. asthma) that are on the dose of more than 400 micro gram/day of budesonide or equivalents inhaled for longer than 1 month during a year,
* Poorly controlled pituitary insufficiencies of other axes (e.g., thyroid-stimulating hormone, adrenocorticotropic hormone/cortisol, vasopressin-deficiency), Major medical conditions and/or presence of contraindication to rhGH treatment.
* Known or suspected HIV-positive patient or patient with advanced diseases such as AIDS or tuberculosis, Drug, substance, or alcohol abuse, Known hypersensitivity to the components of study medication, Evidence of tumour growth or malignant disease in remission for less than one year At screening, presence of anti-hGH antibodies
* The patient and/or the parent/legal guardian are likely to be non-compliant in respect to study conduct.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2003-06; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Annualised HV after 12/24 months treatment and HV SDS height velocity | 12/24 months

SECONDARY OUTCOMES:
HVSDS, HTG, HTSD, bone maturation (BM), IGF-I, IGFBP-3 | 12/24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ference Peter, MD, Principal Investigator — BUDA Children's Hospital, Budapest